CLINICAL TRIAL: NCT05273502
Title: Characterization, Creativity, Leadership, and Search for Solutions to Improve the Lifestyles of Earlier Elderly People in Rural Areas
Brief Title: Earlier Elderly People in Rural Areas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Rosa Sola, MD, PhD. Full professor, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Earlier-Elderly Rural People
Record Dates: First submitted 2022-02-17; First posted 2022-03-10 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Health Behavior; Sarcopenia; Nutrition; Sleep; Physical Activity; Lifestyle, Healthy
MeSH Terms: conditions — Health Behavior; Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (cluster)
Who Masked: Outcomes Assessor
Masking Description: This is an educational program, so that, the intervention group will know that will receive some educational and behavioral activities, and the control group will know that they will not receive any kind of activities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citizen Science Behavioral Intervention (Experimental): The intervention group (IG) participants will receive the whole citizen science intervention of the project, and participants will be assessed at baseline and end-of-study.
  Interventions: Behavioral: Citizen Science intervention
- Control group (No Intervention): The controls group (CG) participants will not receive any kind of intervention, and participants will only be assessed at baseline and end-of-study.

INTERVENTIONS:
Behavioral: Citizen Science intervention — Intervention generated by a participatory research process (co-creation) in the elderly population living in rural areas to co-create solutions to improve their lifestyles, quality of life and health.
  Arms: Citizen Science Behavioral Intervention

SUMMARY:
Social innovation in aging needs to bring new ideas and services to meet new social and welfare needs identified in recent years. In our environment, people ≥60 years old accounted for 20% -24% of the population in 2015, and it is expected to increase to ≥30% by 2050. Older people living in rural areas have been severely affected by confinement, and new needs are being generated. To better understand the needs, an innovative element of this project is to involve the elderly-young people (60-74 years) from rural areas in the generation of solutions, which will make these solutions especially adapted to their needs. It also aims to study the effectiveness of a health education intervention based on participatory research, where young seniors co-create and implement the intervention among their peers, and focused on improving lifestyles, to prevent or to improve sarcopenia.

The objectives of this project are: To characterize the elderly (60 to 74 years) who live independently in rural areas of the province of Tarragona, to actively involve them, through a process of participatory research to generate solutions.

To achieve this goal, it is proposed to make a diagnosis of their health status (lifestyles, risk of malnutrition and sarcopenia), and conduct group interviews (focus groups) including earlier elderly people from rural areas. In addition, participants will receive the intervention co-created by themselves, and the effectiveness of the intervention created will be evaluated.

DETAILED DESCRIPTION:
Social innovation in aging needs to bring new ideas and services to meet new social and welfare needs identified in recent years. In our environment, people ≥60 years old accounted for 20% -24% of the population in 2015, and it is expected to increase to ≥30% by 2050. For the first time in history, most people can aspire to live well beyond the age of 60. On the other hand, the Covid-19 pandemic has severely affected people ≥60 years of age, and may make the welfare and health problems of this population more evident, such as unhealthy lifestyles, the risk of malnutrition, and sarcopenia (defined as loss of muscle mass, strength, and function), which leads to significant dependency and quality of life problems. In addition, older people living in rural areas have been severely affected by confinement, and new needs are being generated. To better understand the needs, an innovative element of this project is to involve the elderly-young people (60-74 years) from rural areas in the generation of solutions, which will make these solutions especially adapted to their needs. Therefore increase the adherence to the solutions created, and also the long-term sustainability of the solutions. It also aims to study the effectiveness of a health education intervention based on participatory research, where young seniors co-create and implement the intervention among their peers, and focused on improving lifestyles, to prevent or to improve sarcopenia.

The objectives of this project are: To characterize the elderly (60 to 74 years) who live independently in rural areas of the province of Tarragona, to actively involve them, through a process of participatory research to generate solutions.

To achieve this goal, it is proposed to make a diagnosis of their health status (lifestyles, risk of malnutrition and sarcopenia), and conduct group interviews (focus groups) including earlier elderly people from rural areas, and the sectors involved, to determine their needs, interests, and barriers to pursuing healthy lifestyles. Based on the information obtained in the diagnosis and group interviews, there will be processes for co-creating solutions based on proposed activities or changes in their immediate environment. During the co-creation process, the elderly and the sectors involved in the 4-helix (government, industry, university, and civil society) will be involved. In addition, participants will receive the intervention co-created by themselves, and the effectiveness of the intervention created will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* People ≥60 years and ≤74 years,
* That they have informed consent,
* Living at home (living independently), Community-dwelling early-elderly
* That they can continue the study,
* They live in the province of Tarragona.

Exclusion Criteria:

* Failure to comply with the inclusion criteria will be considered an exclusion criterion.

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Risk of sarcopenia (muscle strength) | Baseline and through study completion, an average of 1 year
  Change of muscle strength: <27kg in men and <16kg in women measured by a dynamometer
Diagnosis of sarcopenia (muscle strength) | Baseline and through study completion, an average of 1 year
  Change of muscle strength (<27kg in men and <16kg in women measured by a dynamometer)
Diagnosis of sarcopenia (muscle mass) | Baseline and through study completion, an average of 1 year
  Change of muscle mass (<20kg in men and <15kg in women measured by bioimpedance)
Diagnosis of severe sarcopenia (muscle strength) | Baseline and through study completion, an average of 1 year
  Change of muscle strength (<27kg in men and <16kg in women measured by a dynamometer)
Diagnosis of severe sarcopenia (muscle mass) | Baseline and through study completion, an average of 1 year
  Change of muscle mass (<20kg in men and <15kg in women measured by bioimpedance)
Diagnosis of severe sarcopenia (muscle function) | Baseline and through study completion, an average of 1 year
  Change of muscle function (≤0.8 m / s)

SECONDARY OUTCOMES:
Nutrition | Baseline and through study completion, an average of 1 year
  Food frequency questionnaire (not scale)
Physical activity | Baseline and through study completion, an average of 1 year
  International physical activity questionnaire for elderly
  * Low category: non-physical activity or it is not enough to achieve moderate or high category
  * Moderate category: 3 or more days / weeks (vigorous physical activity, at least 25 minutes/day), or 5 or more (moderate physical activity, at least 30 minutes/day), or 5 or more days / weeks of a combination of walking, or moderate-vigorous physical activity (at least 600 METS).
  * High category: 7 or more days / week of a combination of walking, or moderate-vigorous physical activity (at least 3000 METS).
Sleep behaviour | Baseline and through study completion, an average of 1 year
  Pittsburg questionnaire The questionnaire contains a total of 19 questions, grouped into 10 questions. The 19 questions are combined to form seven areas with their corresponding score, each of which shows a range between 0 and 3 points. In all cases, a score of "0" indicates ease, while a score of 3 indicates severe difficulty, within their respective area. The score of the seven areas is finally added to give an overall score, which ranges from 0 to 21 points. "0" indicates ease of sleeping and "21" severe difficulty in all areas.
Risk of malnutrition | Baseline and through study completion, an average of 1 year
  Mini Nutritional Assessment
  12-14 points: normal nutritional status 8-11 points: risk of malnutrition 0-7 points: malnutrition
Weight | Baseline and through study completion, an average of 1 year
  Weight using a balance
height | Baseline and through study completion, an average of 1 year
  Height using a tallimeter

OTHER OUTCOMES:
Age | Baseline and through study completion, an average of 1 year
  Age in years
Gender | Baseline
  Female or male

CONTACTS AND LOCATIONS:
Locations (1):
- University Rovira i Virgili, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No